CLINICAL TRIAL: NCT00333723
Title: A 24-Week Randomized, Double-blind Study to Evaluate the Efficacy, Safety and Tolerability of AVANDIA (8mg Once Daily) in Combination With Glyburide in African American and Hispanic Patients With Type 2 Diabetes Mellitus Who Are Inadequately Controlled on Glyburide Monotherapy
Brief Title: AVANDIA With Glyburide In African American And Hispanic Patients With Type 2 Diabetes Not Controlled by Glyburide Alone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 49653/143
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Rosiglitazone; Glyburide; Type 2 Diabetes Mellitus; African American; Hispanic
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rosiglitazone

SUMMARY:
This study was designed to evaluate the safety and efficacy of AVANDIA (rosiglitazone) (8mg once daily) in African American and Hispanic patients with type 2 diabetes mellitus. As microvascular and macrovascular disease are significant contributors to diabetes morbidity and mortality and previous studies suggest that the thiazolidinedione compounds could have potentially beneficial vascular effects, the effects of rosiglitazone therapy on serum parameters associated with endothelial dysfunction, vascular inflammation and impaired fibrinolysis were examined in this study. Improvement in these parameters suggests that rosiglitazone may provide an additional beneficial vascular effect, apart from its ability to improve glycemic control.

ELIGIBILITY:
Inclusion criteria:

* African American or Hispanic.
* Type 2 diabetes mellitus.
* FPG>=140mg/dL plus HbA1c>=7.5% whilst receiving SU monotherapy.

Exclusion criteria:

* Patients who use insulin.
* Clinically significant liver, kidney or heart disease, including high blood pressure.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2000-07-28 (Actual); Primary Completion 2003-01-06 (Actual); Study Completion 2003-01-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of rosiglitazone combined with glyburide to glyburide monotherapy in reducing glycosylated hemoglobin (HbA1c). | 24 Weeks

SECONDARY OUTCOMES:
Efficacy of rosiglitazone combined with glyburide to glyburide monotherapy upon FPG, c-peptide, HOMA and responder rates. | 24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Abstract: Rosiglitazone Added to Sulfonylurea Improves Glycemic Control and Insulin Sensitivity in African American and Hispanic American Subjects with Type 2 Diabetes, CAMPBELL, JOHN C.; GOULD, ERROL M.; WATERHOUSE, BRIAN R.; COBITZ, ALEXANDER R. Orlando, FL; USA. 64th Annual Scientific Sessions of the American Diabetes Association. 6/4/2004
- [Result] Campbell JC, Gould EM, Waterhouse BR, Cobitz AR. Rosiglitazone added to sulfonylurea improves glycemic control and insulin sensitivity in African American and Hispanic American subjects with type 2 diabetes. Diabetes 2004;53(Suppl 2):A154. Poster 645 presented at ADA.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 49653/143 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 49653/143 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 49653/143 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 49653/143 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 49653/143 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 49653/143 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 49653/143 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register